CLINICAL TRIAL: NCT04887922
Title: The Effect of Preoperative and Postoperative Incentive Spirometry in Patients Undergoing Major Abdominal Surgery
Brief Title: Preoperative and Postoperative Incentive Spirometry in Patients Undergoing Major Abdominal Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Feasibility issues
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 202105028
Record Dates: First submitted 2021-05-10; First posted 2021-05-14 (Actual); Results first posted 2023-05-17 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-04

CONDITIONS: Abdominal Surgery

STUDY DESIGN:
Intervention Model Description: * Prior to surgery, participants will be randomized into three groups: (1) control group with no IS, (2) standard IS, and (3) digital IS + text message.
  * Following surgery, patients will be re-randomized into two groups: (1) standard IS, and (2) digital IS + text message.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (5):
- Pre-Surgery: No Incentive Spirometry (IS) (No Intervention): -Will not receive a incentive spirometer prior to surgery
- Pre-Surgery: Standard Incentive Spirometry (IS) (Experimental): * Will receive a conventional spirometer prior to surgery
  * Will be asked to perform spirometry 30 times per day.
  Interventions: Device: Conventional spirometer
- Pre-Surgery: Digital Incentive Spirometry (IS) + Text Message (Experimental): * Will receive the digital incentive spirometer (Spirobank G) that is compatible with health monitoring software developed by ZEPHYRx®. The digital spirometer couples with a HIPAA-compliant mobile application that calculates and stores pulmonary function test (PFT) results.
  * Will be asked to perform spirometry 10 times per hour, every hour while awake, every day for at least 7 days prior to surgery. Absence of spirometry for 24 hours will trigger a text message reminder to encourage compliance with IS.
  Interventions: Device: MIR Spirobank G; Device: ZEPHYRx®
- Post-Surgery: Standard Incentive Spirometry (IS) (Active Comparator): * After surgery, the participants will receive a conventional spirometer.
  * Will be instructed to perform spirometry 10 times per hour, every hour while awake through postoperative Day 3
  * The conventional spirometer will be equipped with an accelerometer that will allow the research team to determine whether the spirometer moves throughout the patients' postoperative stay (as a proxy for IS use)
  Interventions: Device: Conventional spirometer
- Post-Surgery: Digital Incentive Spirometry (IS) + Text Message (Experimental): * After surgery, the participants will receive the digital incentive spirometer (Spirobank G) that is compatible with health monitoring software developed by ZEPHYRx®. The digital spirometer couples with a HIPAA-compliant mobile application that calculates and stores pulmonary function test (PFT) results.
  * Will be instructed to perform spirometry 10 times per hour, every hour while awake through postoperative Day 3
  * Will receive text reminders to perform spirometry if they do not perform spirometry in a 24-hour period.
  Interventions: Device: MIR Spirobank G; Device: ZEPHYRx®

INTERVENTIONS:
Device: MIR Spirobank G — FDA-approved, Bluetooth digital spirometer
  Arms: Post-Surgery: Digital Incentive Spirometry (IS) + Text Message; Pre-Surgery: Digital Incentive Spirometry (IS) + Text Message
Device: ZEPHYRx® — ZEPHYRx® has developed a 1) digital Bluetooth-enabled IS that allows for the continuous and objective remote monitoring of patient compliance with pre- and postoperative IS via a smartphone app and online provider dashboard.
  Arms: Post-Surgery: Digital Incentive Spirometry (IS) + Text Message; Pre-Surgery: Digital Incentive Spirometry (IS) + Text Message
Device: Conventional spirometer — Will be provided to participants
  Arms: Post-Surgery: Standard Incentive Spirometry (IS); Pre-Surgery: Standard Incentive Spirometry (IS)

SUMMARY:
The goal of this study is to determine the efficacy of incentive spirometry (IS) to improve pulmonary function in the preoperative and postoperative surgical setting. The investigators hypothesize that IS will improve pulmonary function for patients undergoing major abdominal surgery when controlling for protocol compliance. Additionally, the investigators hypothesize that a digital IS device enabled with a text message-based mobile health intervention will improve pulmonary pre-habilitation and rehabilitation, as well as postoperative compliance with the IS device.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo major abdominal surgery with expected postoperative length of stay of 48 hours or more.
* Access to a smartphone.
* At least 18 years of age.
* Ability to understand and willingness to sign an IRB approved written informed consent document.

Exclusion Criteria:

* Younger than 18 years of age
* No access to a smartphone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2022-05-03 (Actual); Primary Completion 2022-12-27 (Actual); Study Completion 2022-12-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chet Hammill, M.D., MCR, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Period: 1st Randomization
Arm/Group | Pre-Surgery: No Incentive Spirometry (IS) | Pre-Surgery: Standard Incentive Spirometry (IS) | Pre-Surgery: Digital Incentive Spirometry (IS) + Text Message | Post-Surgery: Standard Incentive Spirometry (IS) | Post-Surgery: Digital Incentive Spirometry (IS) + Text Message
Started | 1 | 1 | 0 | 0 | 0
Completed | 1 | 0 | 0 | 0 | 0
Not Completed | 0 | 1 | 0 | 0 | 0
Not completed — Decided not to have surgery | 0 | 1 | 0 | 0 | 0
Period: 2nd Randomization
Arm/Group | Pre-Surgery: No Incentive Spirometry (IS) | Pre-Surgery: Standard Incentive Spirometry (IS) | Pre-Surgery: Digital Incentive Spirometry (IS) + Text Message | Post-Surgery: Standard Incentive Spirometry (IS) | Post-Surgery: Digital Incentive Spirometry (IS) + Text Message
Started | 0 | 0 | 0 | 0 | 1
Completed | 0 | 0 | 0 | 0 | 1
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Only 2 participants were enrolled to the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pre-Surgery: No Incentive Spirometry (IS) | Pre-Surgery: Standard Incentive Spirometry (IS) | Pre-Surgery: Digital Incentive Spirometry (IS) + Text Message | Post-Surgery: Standard Incentive Spirometry (IS) | Post-Surgery: Digital Incentive Spirometry (IS) + Text Message | Total
Number analyzed (Participants) | 1 | 1 | 0 | 0 | 0 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 |  |  |  | 0
  Between 18 and 65 years | 1 | 0 |  |  |  | 1
  >=65 years | 0 | 1 |  |  |  | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 |  |  |  | 1
  Male | 0 | 1 |  |  |  | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 |  |  |  | 0
  Not Hispanic or Latino | 1 | 1 |  |  |  | 2
  Unknown or Not Reported | 0 | 0 |  |  |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 |  |  |  | 0
  Asian | 0 | 0 |  |  |  | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 |  |  |  | 0
  Black or African American | 1 | 0 |  |  |  | 1
  White | 0 | 1 |  |  |  | 1
  More than one race | 0 | 0 |  |  |  | 0
  Unknown or Not Reported | 0 | 0 |  |  |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 |  |  |  | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Forced Expiratory Volume in One Second Parameter (FEV1)
Time Frame: From baseline to day-of-surgery preoperative
Population: The participant in the Pre-Surgery: Standard Incentive Spirometry arm only had baseline data available.
Measure: Number; unit: L
Arm/Group | Pre-Surgery: No Incentive Spirometry (IS) | Pre-Surgery: Standard Incentive Spirometry (IS)
Number analyzed (Participants) | 1 | 1
L
  Baseline | 2.42 | 4.07
  Day-of-surgery preoperative: number analyzed (Participants) | 1 | 0
  Day-of-surgery preoperative | 2.46 |

2. Secondary Outcome: Change in Forced Vital Capacity (FVC)
Time Frame: From baseline to day-of-surgery preoperative
Population: The participant in the Pre-Surgery: Standard Incentive Spirometry arm only had baseline data available.
Measure: Number; unit: L
Arm/Group | Pre-Surgery: No Incentive Spirometry (IS) | Pre-Surgery: Standard Incentive Spirometry (IS)
Number analyzed (Participants) | 1 | 1
L
  Baseline | 3.43 | 4.55
  Day-of-surgery preoperative: number analyzed (Participants) | 1 | 0
  Day-of-surgery preoperative | 3.23 |

3. Secondary Outcome: Change in Pulse Oximetry
Time Frame: From baseline to day-of-surgery preoperative
Population: The participant in the Pre-Surgery: Standard Incentive Spirometry arm only had baseline data available.
Measure: Number; unit: percentage of oxygen
Arm/Group | Pre-Surgery: No Incentive Spirometry (IS) | Pre-Surgery: Standard Incentive Spirometry (IS)
Number analyzed (Participants) | 1 | 1
percentage of oxygen
  Baseline | 99 | 97
  Day-of-surgery preoperative: number analyzed (Participants) | 1 | 0
  Day-of-surgery preoperative | 98 |

4. Secondary Outcome: Change in Forced Expiratory Volume in One Second Parameter (FEV1)
Time Frame: From day 1 to postoperative day 3
Population: Only 1 participant is evaluable for this outcome measure as the other enrolled participant did not receive surgery.
Measure: Number; unit: L
Arm/Group | Post-Surgery: Digital Incentive Spirometry (IS) + Text Message
Number analyzed (Participants) | 1
L
  Day 1 | 0.58
  Day 3 | 1.08

5. Secondary Outcome: Change in Forced Vital Capacity (FVC)
Time Frame: From day 1 to postoperative day 3
Population: Only 1 participant is evaluable for this outcome measure as the other enrolled participant did not receive surgery.
Measure: Number; unit: L
Arm/Group | Post-Surgery: Digital Incentive Spirometry (IS) + Text Message
Number analyzed (Participants) | 1
L
  Day 1 | 1.59
  Day 3 | 2.09

6. Secondary Outcome: Change in Pulse Oximetry
Time Frame: From day 1 to postoperative day 3
Population: Only 1 participant is evaluable for this outcome measure as the other enrolled participant did not receive surgery.
Measure: Number; unit: percentage of oxygen
Arm/Group | Post-Surgery: Digital Incentive Spirometry (IS) + Text Message
Number analyzed (Participants) | 1
percentage of oxygen
  Day 1 | 96
  Day 3 | 98

ADVERSE EVENTS:
Time Frame: Adverse events and all-cause mortality was tracked from start of spirometry intervention through post-operative Day 3 (approximately 1 month).
Description: Only 1 participant was evaluable to be followed for adverse event collection and all-cause mortality collection. This one participant was randomized to the Pre-Surgery: No Incentive Spirometry (IS) arm and then after surgery randomized to the Post Surgery: Digital Incentive Spirometry (IS) + Text Message arm.
Groups:
- Post-Surgery: Digital Incentive Spirometry (IS) + Text Message: After surgery, the participants will receive the digital incentive spirometer (Spirobank G) that is compatible with health monitoring software developed by ZEPHYRx®. The digital spirometer couples with a HIPAA-compliant mobile application that calculates and stores pulmonary function test (PFT) results.
  Will be instructed to perform spirometry 10 times per hour, every hour while awake through postoperative Day 3 Will receive text reminders to perform spirometry if they do not perform spirometry in a 24-hour period.
Arm/Group | Pre-Surgery: No Incentive Spirometry (IS) | Pre-Surgery: Standard Incentive Spirometry (IS) | Post-Surgery: Digital Incentive Spirometry (IS) + Text Message
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/0 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-06): https://cdn.clinicaltrials.gov/large-docs/22/NCT04887922/Prot_SAP_000.pdf